CLINICAL TRIAL: NCT02907541
Title: Evaluation of eLearning of Quality Improvement Methods
Brief Title: Protocol for Evaluation of eLearning of Quality Improvement Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); OCB Media (Unknown)
Responsible Party: Principal Investigator, Vimal Sriram, Learning and Improvement Fellow, Chelsea and Westminster NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QI4U
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Learning; Quality Improvement; eLearning
Keywords: eLearning; Quality Improvement Methods; Knowledge Transfer; Impact of learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- QI4U Group (Experimental): Group 1 - Learners who will learn QI methods using eLearning through QI4U
  Interventions: Other: QI4U learning
- Facilitated Learning Group (Active Comparator): Group 2 - Learners who will learn QI methods by facilitated teaching
  Interventions: Other: Facilitated learning
- QI4U and Facilitated Learning Group (Active Comparator): Group 3 - Learners who will learn QI methods using a combination of QI4U and facilitated teaching
  Interventions: Other: QI4U and Facilitated learning

INTERVENTIONS:
Other: QI4U learning — Learners will have access to 8 QI methods modules on QI4U
  Arms: QI4U Group
Other: Facilitated learning — Learners will have access to quarterly learning events and bespoke training on QI methods through facilitated peer-to-peer learning workshops
  Arms: Facilitated Learning Group
Other: QI4U and Facilitated learning — Learners will have access to the 8 QI modules on QI4U and attend quarterly learning events and bespoke training on QI methods through peer-to-peer learning workshops
  Arms: QI4U and Facilitated Learning Group

SUMMARY:
This study evaluates the use of eLearning of quality improvement methods. Participants who use eLearning only, facilitated learning only and a combination of eLearning and facilitated learning will complete questionnaires and be interviewed to establish the effect of eLearning of quality improvement methods to improve knowledge, change in behaviour and impact on healthcare services for better patient care.

DETAILED DESCRIPTION:
Quality improvement (QI) is an increasingly important element of delivering health care. Learning and feeling confident in using QI methods is an essential part of healthcare practice. eLearning is a cost effective way of capacity building to a large cohort of health care professionals and service users. National Institute of Health Research Collaboration for Leadership in Health Research and Care Northwest London has developed a suite of eLearning modules (QI4U) to support an introductory understanding of technical aspects of QI. This protocol describes a trial to evaluate the experience of learning, knowledge gained, change in behaviour, and impact of eLearning of QI methods.

Participants will belong to one of three Groups of learners over the course of 12 months: learners using only QI4U (group 1); people using only facilitated learning (Group 2); and learners using a combination of QI4U and facilitated learning (Group 3). The Kirkpatrick model will be used to evaluate the learning. The primary outcome of interest will be transfer of knowledge gained from learning into clinical practice for service improvement by individuals (level 3). Secondary outcomes will include reaction or experience of QI4U, knowledge gained, and the results or impact of learning through QI4U on service improvement (levels 1, 2 and 4).

Transfer of knowledge into clinical practice will be assessed by interviews with individual learners. Experience of eLearning and knowledge gained will be assessed using feedback forms, questionnaires, time spent doing QI4U and reflective logs. Impact will be assessed by interviews with organisational leads with a high prevalence of QI4U learners.

This study will provide evidence on the effectiveness of using eLearning as a means for learning QI. It will serve to evaluate learners' experience of using eLearning and the impact of various training methods within the context of learning QI.

ELIGIBILITY:
Inclusion Criteria:

* clinicians, managers, commissioners, service users and carers, and researchers who have an interest in learning QI methods.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Transfer of knowledge of QI method into clinical practice | 6-8 months
  Change in behaviour that is a result of learning of QI methods into service improvement projects

SECONDARY OUTCOMES:
Experience of learning measured using eLearning systems success construct questionnaire | Immediately after learning.
  The investigators will use the eLearning systems success construct questionnaire. This is a 36 item survey questionnaire that includes system quality, user satisfaction, net benefits and information quality. Survey items will be rated using a seven-point Likert scale indicating the degree to which respondents agree or disagree.
Knowledge gained measured through the knowledge of QI methods questionnaire | pre learning, immediately after learning and 6-8 months after learning.
  Knowledge of QI methods will be assessed through a question bank of multiple choice questions, the order of the questions are presented in random and learners' knowledge is scored as a percentage of correct answers.
Impact of QI4U learning | 6-8 months
  Impact of QI4U on QI through interviews with executives from trusts that have large cohorts of learners using QI4U

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Sriram, MSc, Principal Investigator — NIHR CLAHRC NWL
Locations (1):
- Nihr Clahrc Nwl, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Glasziou P, Ogrinc G, Goodman S. Can evidence-based medicine and clinical quality improvement learn from each other? BMJ Qual Saf. 2011 Apr;20 Suppl 1(Suppl_1):i13-17. doi: 10.1136/bmjqs.2010.046524. PMID 21450763
- [Background] Ogrinc G, Headrick LA, Morrison LJ, Foster T. Teaching and assessing resident competence in practice-based learning and improvement. J Gen Intern Med. 2004 May;19(5 Pt 2):496-500. doi: 10.1111/j.1525-1497.2004.30102.x. PMID 15109311
- [Background] Batalden P, Davidoff F. Teaching quality improvement: the devil is in the details. JAMA. 2007 Sep 5;298(9):1059-61. doi: 10.1001/jama.298.9.1059. No abstract available. PMID 17785654
- [Background] Wutoh R, Boren SA, Balas EA. eLearning: a review of Internet-based continuing medical education. J Contin Educ Health Prof. 2004 Winter;24(1):20-30. doi: 10.1002/chp.1340240105. PMID 15069909
- [Background] George PP, Papachristou N, Belisario JM, Wang W, Wark PA, Cotic Z, Rasmussen K, Sluiter R, Riboli-Sasco E, Tudor Car L, Musulanov EM, Molina JA, Heng BH, Zhang Y, Wheeler EL, Al Shorbaji N, Majeed A, Car J. Online eLearning for undergraduates in health professions: A systematic review of the impact on knowledge, skills, attitudes and satisfaction. J Glob Health. 2014 Jun;4(1):010406. doi: 10.7189/jogh.04.010406. PMID 24976965
- [Result] Mann KJ, Craig MS, Moses JM. Quality improvement educational practices in pediatric residency programs: survey of pediatric program directors. Acad Pediatr. 2014 Jan-Feb;14(1):23-8. doi: 10.1016/j.acap.2012.11.003. PMID 24369866
- [Result] Boonyasai RT, Windish DM, Chakraborti C, Feldman LS, Rubin HR, Bass EB. Effectiveness of teaching quality improvement to clinicians: a systematic review. JAMA. 2007 Sep 5;298(9):1023-37. doi: 10.1001/jama.298.9.1023. PMID 17785647
- [Result] Wong BM, Etchells EE, Kuper A, Levinson W, Shojania KG. Teaching quality improvement and patient safety to trainees: a systematic review. Acad Med. 2010 Sep;85(9):1425-39. doi: 10.1097/ACM.0b013e3181e2d0c6. PMID 20543652
- [Result] Singh MK, Ogrinc G, Cox KR, Dolansky M, Brandt J, Morrison LJ, Harwood B, Petroski G, West A, Headrick LA. The Quality Improvement Knowledge Application Tool Revised (QIKAT-R). Acad Med. 2014 Oct;89(10):1386-91. doi: 10.1097/ACM.0000000000000456. PMID 25119555
- [Result] Wang Y-S, Wang H-Y, Shee DY. Measuring e-learning systems success in an organizational context: Scale development and validation. Comput. Human Behav. 2007;23:1792-808.
- See also: QI4U website — http://qi4u.ocbmedia.com/login
- See also: Mapping research capacity activities in the CLAHRC community report — https://drive.google.com/file/d/0B7Zq0J4mkDqeWDRQbGRlUlZudWc/view?pref=2&pli=1